CLINICAL TRIAL: NCT05036512
Title: A Double-Blind, Randomized, Placebo-Controlled, Single and Multiple Ascending Dose (SAD/MAD) Study to Evaluate the Safety, Tolerability, PK, and Food Effect of GBT021601, a Hemoglobin S Polymerization Inhibitor, in Healthy Participants.
Brief Title: A Study to Evaluate GBT021601 in Single and Multiple Doses in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBT021601-011; C5351001 (Other: Pfizer)
Record Dates: First submitted 2021-08-13; First posted 2021-09-05 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo as a tablet or capsule with dose based off of preceding cohort's data.
  Interventions: Drug: GBT021601
- GBT021601 (Experimental): GBT021601 as a tablet or capsule with dose based off of preceding cohort's data.
  Interventions: Drug: GBT021601

INTERVENTIONS:
Drug: GBT021601 — Administered orally with water as a single dose in the morning.
  Other Names: Placebo

SUMMARY:
This first in human study is designed to evaluate the safety, tolerability, pharmacokinetics (PK), and food effect of GBT021601, a hemoglobin S (HbS) polymerization inhibitor, in healthy participants.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, single and multiple ascending dose study in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females ≥ 18 to ≤ 55 years of age
* Body mass index ≥ 18.0 to ≤ 30.0 kg/m2
* Body weight ≥ 50 kg at screening and Day -1

Exclusion Criteria:

- Positive pregnancy test or currently breastfeeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Safety, as assessed by frequency and severity of adverse events (AEs) | 119 days from screening Part A, 134 days from screening Part B
  AEs will be coded to system organ class and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA) and summarized.
Safety, as assessed by changes in Heart Rate. | 119 days from screening Part A, 134 days from screening Part B
  Number of participants with changes in heart rate (bpm) as compared to baseline.
Safety, as assessed by changes in eGFR | 119 days from screening Part A, 134 days from screening Part B
  Number of participants with changes in eGFR from baseline
Safety, as assessed by changes in alanine aminotransferase (ALT) | 119 days from screening Part A, 134 days from screening Part B
  Number of participants with changes in alanine aminotransferase (ALT)
Safety, as assessed by changes in Blood pressure | 119 days from screening Part A, 134 days from screening Part B
  Number of participants with changes in systolic (mmHg) and diastolic (mmHg) blood
Plasma concentration | 119 days from screening Part A
  Time of Cmax
Plasma concentration | 134 days from screening Part B
  Cmax on D1-D15

SECONDARY OUTCOMES:
Determine whole blood concentration of GBT021601 | 119 days from screening Part A
  Hemoximetry will be used to assess oxygen saturation in whole blood by generating oxygen equilibrium curves (OECs) which relate the extent of Hb-O2 saturation to the partial pressure of O2 (pO2) and measure the binding affinity of O2 to Hb.
Determine plasma concentration of GBT021601. | 134 days from screening Part B
  With dosing data from each cohort determine the steady-state maximum plasma/whole blood concentration (Cmax).
Safety, as assessed by changes in QTcF | 119 days from screening Part A, 134 days from screening Part B
  Number of participants with changes in the QTcF interval from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- ICON Early Phase Services, LLC, San Antonio, Texas, United States
- Australia (3):
  - Harry Perkins Institute of Medical Research, Nedlands, Western Australia
  - Linear Clinical Research, Nedlands, Western Australia
  - Oxford Compounding, North Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT021601-011